CLINICAL TRIAL: NCT05314972
Title: Assessment of Foot Alignment and Pressure After Correction of Varus Knee by High Tibial Osteotomy or Total Knee Replacement
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrhman Abdelaziz Khalaf Mohamed, principal investigator, Assiut University
Other Study IDs: foot alignment and pressure
Record Dates: First submitted 2021-12-31; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Varus Deformity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluated the change in foot alignment after TKA or HTO by prospectively analyzing the correlation between the knee joint and the foot deformity, the post-operative improvement in the foot deformity, and the long-term post-operative changes in foot alignment.

DETAILED DESCRIPTION:
The mechanical alignment of the lower extremity is an important consideration in the long-term outcome following total knee arthroplasty (TKA) or high tibial osteotomy (HTO) . Alignment between the hip and the ankle through the knee joint has been used in determining coronal alignment, based on the assumption that weight-bearing forces pass through the centre of the knee joint during neutral mechanical. However, the weight-bearing vector can be affected by hindfoot and midfoot alignment because load is transmitted not from the ankle joint, but from the ground reaction point. Thus hindfoot alignment after knee correction may critically affect the longevity of the prosthesis

Most patients with some degree of knee joint deformity, which in turn may be associated with a deformity of the foot. In fact, an association between varus alignment of the knee joint and valgus alignment of the foot in osteoarthritis patients has been reported. Because the subtalar joint compensates for the knee joint deformity , correction of the deformity after TKA or HTO can affect foot alignment. Improvements in midfoot and hindfoot alignment have been noted in patients with osteoarthritis after correction of deformity. However, foot valgus may also persist, with little improvement after knee correction.

ELIGIBILITY:
Inclusion Criteria:

* all varus aligned knee admitted to Assiut University Hospitals (Total Knee Arthroplasty or High Tibial Osteotomy) .

Exclusion Criteria:

* patient with prior surgery of knee or foot . -secondary osteoarthritis. -valgus knee.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: total coverage of all cases admitted to Assiut University Hospitals in one year
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
: Radiological changes in hindfoot and midfoot alignment after correction of varus knee by High tibial osteotomy (HTO) or total knee arthroplasty(TKA) | 6-12 months
  This study evaluated the change in foot alignment after TKA or HTO by:
  1. prospectively analyzing the correlation between the knee joint and the foot deformity.
  2. post-operative improvement in the foot deformity.
  3. the long-term post-operative changes in foot alignment.

SECONDARY OUTCOMES:
clinical assessment of the foot by american orthopedic foot&ankle society ( AOFAS) before and after knee correction | 6-12 months
  AOFAS covers four different regions of the foot: The ankle-hindfoot, midfoot, metatarsophalangeal (MTP)-interphalangeal (IP) for the hallux, and MTP-IP for the lesser toes.These four anatomic regions have their own version of the AOFAS survey. Each c is designed to be used independent of the others. However, each measure is comprised of nine questions and cover three categories: Pain (40 points), function (50 points) and alignment (10 points). These are all scored together for a total of 100 points

REFERENCES:
- [Background] Bargren JH, Blaha JD, Freeman MA. Alignment in total knee arthroplasty. Correlated biomechanical and clinical observations. Clin Orthop Relat Res. 1983 Mar;(173):178-83. PMID 6825330
- [Background] Fang DM, Ritter MA, Davis KE. Coronal alignment in total knee arthroplasty: just how important is it? J Arthroplasty. 2009 Sep;24(6 Suppl):39-43. doi: 10.1016/j.arth.2009.04.034. Epub 2009 Jun 24. PMID 19553073
- [Background] Jeffery RS, Morris RW, Denham RA. Coronal alignment after total knee replacement. J Bone Joint Surg Br. 1991 Sep;73(5):709-14. doi: 10.1302/0301-620X.73B5.1894655.
- [Background] Longstaff LM, Sloan K, Stamp N, Scaddan M, Beaver R. Good alignment after total knee arthroplasty leads to faster rehabilitation and better function. J Arthroplasty. 2009 Jun;24(4):570-8. doi: 10.1016/j.arth.2008.03.002. Epub 2008 May 19. PMID 18534396
- [Background] Cho WS, Cho HS, Byun SE. Changes in hindfoot alignment after total knee arthroplasty in knee osteoarthritic patients with varus deformity. Knee Surg Sports Traumatol Arthrosc. 2017 Nov;25(11):3596-3604. doi: 10.1007/s00167-016-4278-8. Epub 2016 Aug 16. PMID 27527338
- [Background] Norton AA, Callaghan JJ, Amendola A, Phisitkul P, Wongsak S, Liu SS, Fruehling-Wall C. Correlation of knee and hindfoot deformities in advanced knee OA: compensatory hindfoot alignment and where it occurs. Clin Orthop Relat Res. 2015 Jan;473(1):166-74. doi: 10.1007/s11999-014-3801-9. PMID 25024033
- [Background] Hara Y, Ikoma K, Arai Y, Ohashi S, Maki M, Kubo T. Alteration of hindfoot alignment after total knee arthroplasty using a novel hindfoot alignment view. J Arthroplasty. 2015 Jan;30(1):126-9. doi: 10.1016/j.arth.2014.07.026. Epub 2014 Jul 25. PMID 25155238
- [Background] Mullaji A, Shetty GM. Persistent hindfoot valgus causes lateral deviation of weightbearing axis after total knee arthroplasty. Clin Orthop Relat Res. 2011 Apr;469(4):1154-60. doi: 10.1007/s11999-010-1703-z. Epub 2010 Dec 1. PMID 21120711